CLINICAL TRIAL: NCT06727396
Title: A Phase 1, Randomized, Double-Blinded, Placebo-Controlled, Parallel-Group, Single Center Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of CKD-508 in Healthy Participants.
Brief Title: A Study to Investigate the Safety, Tolerability, PK, and PD of CKD-508 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A104_02PK2405
Record Dates: First submitted 2024-12-02; First posted 2024-12-10 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- CKD-508 dose level 1 (Experimental): Multiple dose of CKD-508 tablets
  Interventions: Drug: CKD-508 Tablet
- CKD-508 dose level 2 (Experimental): Multiple dose of CKD-508 tablets
  Interventions: Drug: CKD-508 Tablet
- CKD-508 dose level 3 (Experimental): Multiple dose of CKD-508 tablets
  Interventions: Drug: CKD-508 Tablet
- CKD-508 dose level 4 (Experimental): Multiple dose of CKD-508 tablets
  Interventions: Drug: CKD-508 Tablet
- Placebo (Placebo Comparator): Multiple dose of placebo tablets
  Interventions: Drug: Placebo Tablet

INTERVENTIONS:
Drug: CKD-508 Tablet — Investigational drug
  Arms: CKD-508 dose level 1; CKD-508 dose level 2; CKD-508 dose level 3; CKD-508 dose level 4
Drug: Placebo Tablet — Placebo
  Arms: Placebo

SUMMARY:
This Phase 1, randomized, parallel-group, placebo-controlled, double-blinded study aims to evaluate the safety, PK, and PD of CKD-508 when administered multiple times once daily to healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* The participant is capable of providing signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and the protocol.
* Male and female adults aged 18 to 55 years at screening.
* Healthy participants were determined by pre-study medical evaluation and judged by the Investigator.
* Female participants of non-childbearing potential (surgically sterile [hysterectomy or oophorectomy]) or postmenopausal (amenorrhea for more than 12 months with follicle-stimulating hormone [FSH] in the postmenopausal range as confirmed by an FSH test).
* Female participants of childbearing potential who agree to use highly effective method of contraception in the protocol consistently and correctly from screening until the last dose administration of the study intervention.
* Male participants must be unable to procreate (defined as surgically sterile [had a vasectomy] ≥6 months prior screening) or must agree to use a highly effective contraception as detailed in the protocol during the intervention period and for at least 90 days after the study completion and refrain from donating sperm during this period.
* Non-smoker (or other nicotine use) as determined by history (no nicotine use over the past 6 months) and by urine cotinine concentration (<200 ng/mL) at screening and admission.

Exclusion Criteria:

* History or evidence of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological, or psychiatric disorder as determined by the Investigator.
* Presence of any disorder that would interfere with the absorption, distribution, metabolism, or excretion of study intervention as judged by the Investigator.
* Serum alkaline phosphatase (ALP) or total bilirubin ≥upper limit of normal (ULN), or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >ULN at either screening or admission.
* Abnormal renal function with estimated glomerular filtration rate (eGFR) <90 mL/min/1.73 m2 at screening.
* History or presence of clinically significant abnormal cardiac automaticity, heart rhythm, ECG findings, or other relevant conditions that may pose a risk to the participants as judged by the Investigator.
* History of alcohol and/or illicit drug abuse within 2 years before screening or positive urine test for alcohol or positive urine drug test at screening or admission.
* Positive test for HBsAg, HCV RNA, or HIV antibody at screening.
* Currently taking a lipid-modifying medication.
* History of hypersensitivity to CKD-508 or medicinal products with similar chemical structures.
* Individual unlikely to comply with the protocol requirements, instructions, and study-related restrictions.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience a Treatment-Emergent Adverse Event (TEAE) | up to Day 56
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. A TEAE will be defined as any AE that emerges during treatment (i.e., AE which starts during or after study drug administration or pre-existed and worsened in severity after study drug administration), and those will be analyzed for the purpose of safety analysis. The number of participants who experience a TEAE will be reported.
Maximum Plasma Concentrations of CKD-508 after single and multiple doses | up to Day 56
  Peak plasma concentration (Cmax)
Time to Maximum Plasma Concentrations of CKD-508 after single and multiple doses | up to Day 56
  Time of peak plasma concentration (Tmax)
Area Under the Concentration-Time Curve of CKD-508 after single dose | up to 24 hours post-dose
  Area under the concentration-time curve from pre-dose (time 0) to post-dose 24 h (AUC0-24h) after a single dose
Area Under the Concentration-Time Curve of CKD-508 after multiple doses | up to Day 56
  Area under the concentration-time curve from pre-dose (time 0) to post-dose 24 h (AUCtau.ss) after multiple doses
Change from baseline in CETP activity after multiple doses of CKD-508 or placebo | up to Day 56
  The absolute values and percentages of change from baseline in CETP activity measured in blood after multiple doses of CKD-508 or placebo

SECONDARY OUTCOMES:
Change from Baseline in Low-density Lipoprotein Cholesterol (LDL-C) after multiple doses of CKD-508 or placebo | up to Day 40
  The absolute values and percentages of change from baseline in LDL-C measured in blood after multiple doses of CKD-508 or placebo
Change from Baseline in High-density Lipoprotein Cholesterol (HDL-C) after multiple doses of CKD-508 or placebo | up to Day 40
  The absolute values and percentages of change from baseline in HDL-C measured in blood after multiple doses of CKD-508 or placebo
Change from Baseline in CETP mass after multiple doses of CKD-508 or placebo | up to Day 56
  The absolute values and percentages of change from baseline in CETP protein concentration measured in blood after multiple doses of CKD-508 or placebo
The effects on the cardiac repolarization by assessing the QTc interval after single and multiple doses of CKD-508 or placebo | up to Day 56

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Glendale, California, United States